CLINICAL TRIAL: NCT06230354
Title: A RAndomised Placebo Controlled Trial - to Explore the Efficacy and Mechanism of Action of Tezepelumab in Eosinophilic Granulomatosis With Polyangiitis
Brief Title: Explore the Efficacy and Mechanism of Action of Tezepelumab in Eosinophilic Granulomatosis With Polyangiitis
Acronym: RACEMATE
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1007564; 21HH7284 (Other: IMPERIAL)
Record Dates: First submitted 2024-01-08; First posted 2024-01-30 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: EGPA - Eosinophilic Granulomatosis With Polyangiitis
Keywords: EGPA; Eosinophilic granulomatosis with polyangiitis; Tezepelumab; Mechanism; Alarmin; Vasculitis; Experimental Medicine
MeSH Terms: conditions — Churg-Strauss Syndrome; Vasculitis | interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tezepelumab (Experimental): Tezepelumab subcutaneous injection
  Interventions: Drug: Tezepelumab
- Placebo (Placebo Comparator): Placebo subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tezepelumab — Tezepelumab subcutaneous injection
  Arms: Tezepelumab
Drug: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
RACEMATE is a phase 2b, multicentre, randomised, double-blinded, placebo-controlled study designed to explore the efficacy and mechanism of action of tezepelumab in adults with eosinophilic granulomatosis with polyangiitis (EGPA).

DETAILED DESCRIPTION:
RACEMATE is a randomised double-blind placebo-controlled experimental medicine study designed to explore both the efficacy and mechanism of action of tezepelumab (210 milligram [mg] administered subcutaneously [SC] every 4 weeks) compared with placebo over a 24-week study treatment period in subjects with active (non-severe) Eosinophilic Granulomatosis with Polyangiitis (EGPA) receiving standard of care therapy including background corticosteroid therapy with or without immunomodulatory therapy. This study will take place across 16 centres in the United Kingdom. Corticosteroid dose will be tapered during the treatment period in accordance with standard of care.

The key outcome of this study focuses on evaluation of clinical remission, defined as a Birmingham Vasculitis Activity Score (BVAS) version 3 of 0 and receipt of prednisolone ≤ 4mg daily and no receipt of oral corticosteroids above baseline during the treatment period. Secondary outcomes will include reduction in disease flare, improvement in scores for asthma control, sino-nasal disease and spirometry amongst others.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of providing written informed consent
2. Eosinophilic granulomatosis with polyangiitis is defined as a history of asthma, a blood eosinophil level of 10% or an absolute eosinophil count of more than 1.0 x10^9/L, and the presence of two or more criteria:

   - Histopathological evidence of eosinophilic vasculitis

   - Perivascular eosinophilic infiltration, or eosinophil-rich granulomatous inflammation

   - Neuropathy

   - Pulmonary infiltrate
   * Sino-nasal abnormality
   * Cardiomyopathy
   * Glomerulonephritis
   * Alveolar haemorrhage
   * Palpable purpura
   * Anti-neutrophil cytoplasmic antibody [ANCA] positivity
3. History of one or more flares of EGPA in 24 months prior to screening. EGPA flares will be defined as worsening or persistence of active disease characterised by:

   - Active vasculitis (BVAS >0); OR

   - An asthma exacerbation/asthma worsening OR

   - Active nasal and/or sinus disease

   Warranting:

   - Rescue use of prednisolone for 3 or more days OR an increase in background prednisolone dose by at least 5 mg daily for at least three days OR

   - An increased dose or addition of immunosuppressive therapy; OR
   * Hospitalisation related to EGPA worsening
4. Blood eosinophil level at screening (visit 1) of ≥ 0.2 x10^9/L (participants can be re screened once within 2 weeks if the BEC is < 0.2 x10^9/L at the initial screening assessment).

   n.b. This criterion is not relevant for participants taking background anti-IL-5/5R biological agents mepolizumab (MEPO) or benralizumab (BRZ) in which any baseline blood eosinophil count (BEC) permitted.
5. Non severe EGPA according to the American College of Rheumatology 2021 definition.

Non-Severe EGPA: Vasculitis without life- or organ-threatening manifestations (e.g., rhinosinusitis, asthma, mild systemic symptoms, uncomplicated cutaneous disease, mild inflammatory arthritis).

6. Stable dose of prednisolone (≥5.0 to ≤30.0 mg per day, with or without additional Immunomodulatory therapy) for at least 4 weeks before the baseline visit.

7. Immunomodulatory therapy:

(i) If receiving non-biologic immunomodulatory therapy, the dosage must be stable for the 4 weeks prior to baseline visit.

(ii) Patients on background anti-IL-5/5R therapy (either MEPO or BRZ) at any licensed dose for the current clinical indications of severe asthma and EGPA in the UK and Europe respectively AND have been on treatment for at least 6 months.

n.b. participants on background anti-IL-5/5R therapy will be capped to no more than 50% of the total sample size.

Exclusion Criteria:

1. Diagnosis of Granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA).
2. Pregnancy or unable to use a highly effective method of birth control (confirmed by the Investigator) from randomisation throughout the study duration and within 8 weeks after last dose of IMP.
3. Active life- or organ-threatening manifestations of EGPA within 6 months prior to screening, defined as:

   * Severe alveolar haemorrhage
   * Rapidly progressive glomerulonephritis
   * Severe gastrointestinal or central nervous system involvement requiring intensification of immunosuppression or surgery
   * Severe cardiac involvement including life threatening arrhythmia, heart failure with an ejection fraction < 20% or acute myocardial infarction or active myocarditis
4. Current active malignancy.
5. Immunodeficiency including HIV
6. Helminth infection within 6-months of screening that has not been treated or remains refractory to treatment.
7. Unstable liver disease with the exception of Gilberts syndrome or asymptomatic gallstones.
8. Use of a prohibited concurrent medication as listed below:

   * Biologic therapy for severe asthma (except MEPO or BRZ) within 4 months or 5 half-lives (whichever is longer) prior to Visit 1 or receipt of any investigational non-biologic agent within 30 days or 5 half-lives (whichever is longest) prior to Visit 1.
   * Biologic therapies for EGPA including Rituximab and Alemtuzumab within 6 months of visit 1.
   * IV or SC immunoglobulin therapy within 3 months of visit 1.
   * Oral cyclophosphamide within 6 weeks of screening or IV cyclophosphamide within 4 months of visit 1.
   * IM or IV corticosteroids within 6 weeks of visit 1.
9. Known adrenal insufficiency (primary or secondary), that in the opinion of the investigator and clinical care team preclude maintenance oral steroid tapering

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who are in remission at week 24 | Week 24
  The proportion of patients who achieve remission at week 24 (defined as a Birmingham Vasculitis Activity Score (BVAS) version 3 score of 0 and receipt of prednisolone of ≤ 4mg daily and no receipt of oral steroids above baseline dose in the 4 weeks prior to week 24). BVAS is a validated tool for assessment of disease activity in patients with vasculitis with potential scores ranging from 0-63, with higher scores indicating worse disease activity.

SECONDARY OUTCOMES:
Time to first EGPA flare | Up to Week 24
  EGPA flare was defined as worsening or recurrence of active disease since the last visit characterised by active vasculitis (BVAS >0) or active asthma symptoms and/or signs with a corresponding worsening in Asthma Control Questionnaire-6 (ACQ-6) score or active nasal and/or sinus disease, with a corresponding worsening in at least one of the sino-nasal symptom questions warranting: (i) rescue use of prednisolone/equivalent systemic steroid for 3 or more days OR an increase in background prednisolone/equivalent systemic steroid dose by at least 5 mg daily of prednisolone equivalents for at least three days OR (ii) an increased dose or addition of immunosuppressive therapy; OR (iii) hospitalization related to EGPA worsening. The number of participants with at least one EGPA flare during the planned study treatment period are presented.
Total accrued duration of remission | Up to Week 24
  Total accrued weeks of remission defined as defined as a Birmingham Vasculitis Activity Score (BVAS) - version 3, score of 0 with mOCS dose of prednisolone/prednisolone ≤ 4mg/day and BVAS of 0.
Proportion of participants that demonstrate sustained remission | Up to Week 24
  The proportion of patients that demonstrate sustained remission at both weeks 20 and 24 (defined as a BVAS version 3 score of 0 and receipt of prednisolone of ≤ 4 mg daily and no receipt of oral steroids above baseline dose between weeks 16 and 24)
Proportion of participants that tapered mOCS by at least 2.5 mg/day | Up to Week 24
  Proportion of patients that tapered their maintenance oral corticosteroids (mOCS) by at least 2.5 mg/day of prednisolone equivalent during the OCS tapering period, who remained in remission
Change in SinoNasal Outcome Test-22 (SNOT-22) | Between Week 0 and/or Week 12 and Week 24
  Change from baseline (week 0) to weeks 12 & 24 in the SinoNasal Outcome Test-22 questionnaire score (SNOT-22). SNOT-22 is a validated assessment of the burden of chronic rhinosinusitis with potential scores ranging from 0-110, with higher scores indicating a worse impact on health-related quality of life.
Change in European Quality of Life 5 Dimensions 5 Level (EuroQoL-5D-5L) | Up to Week 24
  Change from baseline (week 0) to week 24 in the European Quality of Life 5 Dimensions 5 Level (EuroQoL-5D-5L) questionnaire score. The EuroQoL-5D-5L is a validated standardised descriptive measure of health-related quality of life with potential scores ranging from "no problems" to "extreme problems" in all domains. The questionnaire also asks the participant to indicate their overall health that day on a scale of 0-100, with lower scores indicating worse health.
Change in Juniper 6-item Asthma Control Questionnaire (ACQ-6) | Between Week 0 and/or Week 12 and Week 24
  Change from baseline to week 12 and 24 in Juniper 6-item Asthma Control Questionnaire (ACQ-6) score. The ACQ-6 is a validated assessment of asthma symptom control, with potential scores ranging from 0-6, with higher scores indicating worse asthma symptom control.
Change in blood eosinophil level | Between Week 0 and/or Week 12 and Week 24
  Change from baseline (week 0) to week 12 and 24 in blood eosinophil level
Change in spirometry | Between Week 0 and/or Week 12 and Week 24
  Change from baseline (week 0) to weeks 12 and 24 in pre-bronchodilator FEV1% predicted and FEV1/FVC ratio.
Change in FeNO | Between Week 0 and/or Week 12 and Week 24
  Change from baseline (week 0) to weeks 12 and 24 in Fractional Exhaled Nitric Oxide level (FeNO).
Change in eGFR | Between Week 0 and/or Week 12 and Week 24
  Change from baseline (week 0) to weeks 12 and 24 in estimated glomerular filtration rate (eGFR).

OTHER OUTCOMES:
Glucocorticoid-induced toxic effects | Up to Week 24
  Glucocorticoid-induced toxic effects according to the Glucocorticoid Toxicity Index (GTI) between week 0 and week 24. The GTI provides two GTI scores: the Cumulative Worsening Score (CWS) and the Aggregate Improvement Score (AIS). The GTI-CWS, with potential scores ranging from 0-439, captures cumulative glucocorticoid toxicity regardless of whether it is permanent or transient. The GTI-CWS can only increase or remain the same over time. A higher score indicates higher glucocorticoid toxicity. The GTI-AIS, with potential scores ranging from -346 to +439, captures both worsening and improvement in glucocorticoid toxicity. New or worsening toxicities contribute a positive score and improvement in existing toxicities contributes a negative score. A higher score indicates higher glucocorticoid toxicity.
EGPA flare type | Up to Week 24
  EGPA flare type as assessed by the local investigator according to the following three primary categories: (1) asthma exacerbation, (2) Sino-nasal disease exacerbation, (3) relapse of systemic vasculitis.
Change in nEPX | Between Week 0 and/or Week 12 and Week 24
  Change from baseline (week 0) to weeks 12 and 24 in nasal eosinophil peroxidase (nEPX) level.
Change in uACR | Between Week 0 and/or Week 12 and Week 24
  Change from baseline (week 0) to week 12 and week 24 in urinary albumin to creatinine ratio (uACR).
Change in ANCA | Between Week 0 and/or Week 12 and Week 24
  Change from baseline (week 0) and week 24 in Anti Neutrophil Cytoplasmic Antibody (ANCA) status (defined by immunofluorescence and MPO/PR3 ANCA titres).

CONTACTS AND LOCATIONS:
Overall Officials: Salman Siddiqui, MBBS, Principal Investigator — Imperial College London
Locations (13):
- United Kingdom (13):
  - Aberdeen Royal Infirmary - NHS Grampian, Aberdeen
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University Hospitals of Leicester NHS Trust, Leicester
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust, London
  - Royal Free London NHS Trust, London
  - Guy's Hospital - Guy's and St Thomas' NHS Foundation Trust, London
  - Royal Brompton Hospital - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Foundation Trust, Nottingham
  - University Hospital Southampton NHS Foundation Trust, Southampton